CLINICAL TRIAL: NCT01932983
Title: Clinical Application of Train of Four Testing in the Intraoperative Monitoring Setting
Brief Title: Clinical Application of "Train of Four" Testing in the Intraoperative Monitoring Setting
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S12-01499
Record Dates: First submitted 2013-08-26; First posted 2013-08-30 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Neuromuscular Blockade; Muscle Relaxation
Keywords: Neuromuscular blockade; TOF test; Quantitative TOF method; Visual interpretation of TOF

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TOF test: TOF - train of four test performed on patiens undergoing lumbar spine surgery where introperative neurophysiologic monitoring is applied. Stimulation of peripheral nerve - ulnar nerve resulting with muscle contractions and evaluation of responses by anesthesiologist and neurophysiologists. Stimulation with group of 0.2 millisecond pulses, spaced 500 millisecond apart, at a 2 Hz rate, current 20-60 mA to deliver four muscle contractions. Eligibility criteria included patients for study where subjective visual interpretation and quantitative interpretation of Adductor pollicis muscle responses is followed.
  Interventions: Device: Train of four test

INTERVENTIONS:
Device: Train of four test — TOF test includes stimulation of peripheral nerve of upper extremity, ulnar nerve in this study. Two methods of interpretation are included, visual which uses anesthesiologist TOF device, and quantitative uses intraoperative neurophysiologic monitoring device, both devices are in routine clinical practice use. Different interpretation of muscle contractions are followed, by quantitative method and visual method. Visual evaluates number of twitches and determines the degree of neuromuclular block and percent of blocked acetylcholine receptors. Quantitative method record muscle contraction by using EMG, presents each twitch as amplitude, caluculate peak to peak value, and provide numerical value and difference for each twitch.

SUMMARY:
The study examines the clinical application of TOF (train of four test) used by anesthesiologists and neurophysiologists during instrumented spine procedures, as well as certain associated parameters. 'Train of four' test is a test routinely used during the surgery, which is performed by stimulation of peripheral nerve with purpose to determine the degree of muscle relaxation by interpretation of muscle response. During spine surgery, it is helpful for the surgeon to have a patient's muscles as relaxed as possible with the least amount of tone, especially when exposing. Anesthesiologists achieve this level of relaxation by giving a neuromuscular blocking agent. If medication given to do this has not fully left their system by the time the surgeon needs to start putting in the screws and rods, then the intraoperative monitoring can not be adequately performed. If the muscles are too relaxed, then free run EMG and screw stimulation, two monitoring methods used, will not be analyzed correctly and the surgery may be adversely affected. This study compares the results of the 'train of four' test performed by neurophysiologists and anesthesiologists. Additionally, it looks at the differences, if any, in comparing stimulation of the foot nerve (tibial n.) or hand nerve (ulnar n.) Performing the TOF (train of four test) in the lower extremity can be relevant for many reasons. Train of four tests can show the presence of four twitches in the arms but the legs may not fully recovered from muscle relaxant given by anesthesia. Also, train of four test which uses subjective method of interpretation by anesthesiologists may present different results compared than objective quantitative method of train of four test interpretation. Ultimately, the goal of this study is to show the importance of 'TOF' testing in ensuring that any identifiable preventable intraoperative surgical complication is appropriately identified.

DETAILED DESCRIPTION:
TOF test was performed by two routinely used devices, peripheral nerve stimulator and intraoperative neurophysiologic monitoring device. TOF monitoring of upper extremity included stimulation of ulnar nerve. Negative surface electrode was placed on the wrist in line with the smallest digit 1-2cm below skin crease and the positive 2-3cm proximal to the negative electrode. Active surface recording electrodes were placed on adductor pollicis muscle. TOF monitoring of lower extremity included stimulation of peripheral nerve, posterior tibial nerve. Surface stimulating electrodes were placed, negative over inferolateral aspect of medial malleolus, and positive electrode 2-3cm proximal to the negative electrode. Stimulation current was 20-30 mA for hand and 30-60mA foot TOF by a group of 0.2 millisecond pulses, spaced 500 millisecond apart, to deliver four contractions. Surface recording electrodes were used for measuring muscle response on foot, active electrode which was located on the Flexor hallucis brevis muscle and reference on the big toe. Intraoperative monitoring device was used, and software with TOF monitoring programe was installed. EMG response was calculated by the peak of amplitude (peak to peak amplitude) presented in quantitative value of online measurement. Interpretation was different, visual and subjective. Peripheral nerve stimulator was used for subjective TOF test. Output current was adjustable from 0 to 70 mA. Repeat stimulation of 4 pulses/0.2 milliseconds repeated every 500 milliseconds. Surface negative electrodes were placed over the course of ulnar nerve on the wrist, in line with the smallest digit, 1-2cm proximal from skin crease, and positive electrode 2-3 cm proximal. Response was followed on adductor pollicis muscle. All data were kept in electronic medical records and if data are not complete subjects were not included in the study. Results were compared between TOF methods on two different body sites, upper and lower extremity, by quantitative method and other comparison was made between subjective and quantitative method with TOF test located in both methods on the upper extremity.

ELIGIBILITY:
Inclusion Criteria:

Subject undergoing spine fusion surgery when intraoperative neurophysiologic monitoring is included.

Exclusion Criteria:

Subjects with history of previous nerve injury or peripheral neuropathies when intraoperative neurophysiologic monitoring was precluded. Possible technical issues during surgery prior TOF test such as incorrect electrode placement, lead wire attachment, TOF device error or impossibility to correct it in acceptable time when TOF test can not be performed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing instrumented orthopedic surgical procedure which requires the use of neurophysiologic intraoperative monitoring modalities.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Muscle contraction - TOF twitch after peripheral nerve stimulation | During spine lumbar surgery after pedicle screw placement
  TOF test is performed after pedicle screw placement during lumbar spine surgery, prior neurophysiological pedicle screw position test.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Beric, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, Hospital for Joint Diseases, New York, New York, United States

REFERENCES:
- [Result] Gavrancic B, Lolis A, Beric A. Train-of-four test in intraoperative neurophysiologic monitoring: differences between hand and foot train-of-four. J Clin Neurophysiol. 2014 Dec;31(6):575-9. doi: 10.1097/WNP.0000000000000111. PMID 25462145
- See also: Clinical trial of application of train of four testing in the intraoperative monitoring setting — http://clinicaltrials.gov